CLINICAL TRIAL: NCT00669838
Title: Loco Regional Anesthesia for Dental Treatment in Cardiac Patients: Comparative Study Between Plain Lidocaine 2% and Lidocaine 2% With Epinephrine 1:100.000
Brief Title: Anesthesia for Dental Treatment in Cardiac Patients: Lidocaine Comparative Study
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Joaquim Edson Vieira, Divisão de Anestesia, Hospital das Clínicas da FMUSP
Other Study IDs: CAP432-03
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Arrhythmias; Anxiety
Keywords: Anesthesia, Local; Lidocaine; Dental care; Arrhythmias, Cardiac; Anxiety
MeSH Terms: conditions — Arrhythmias, Cardiac; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PL: Patients who receive local anesthesia with 2% lidocaine without epinephrine
- LE: Patients who receive local anesthesia with 2% lidocaine with 1:100.000 epinephrine

SUMMARY:
Prospective, randomized double-blinded study to investigate hemodynamic changes in valvular cardiac patients during dental treatment with the use of a local anesthesia containing epinephrine.

DETAILED DESCRIPTION:
Patients with valvular disease constitute a group in which local anesthesia must be effective to avoid higher release of endogenous catecholamines that could trigger hemodynamic. The study was conducted in the Dental Department of the Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (Brazil). Patients were allocated into two groups through an aleatory numbered table: PL (plain 2% lidocaine, n= 31) and LE (2% lidocaine with 1:100.000 epinephrine, n= 28). The anesthetic amount was registered. DIXTAL monitor (São Paulo- Brazil) captured blood pressure, heart rate, oxygenation and electrocardiogram records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acquired valvular disease

Exclusion Criteria:

* Patients having platelets counting lower than 70.000 or INR > 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired valvular diseases participated in this study, aging between 18-65 years in need of dental surgery (extractions) or restorative dentistry in mandible
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2003-01; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
arrhythmias | during procedure

SECONDARY OUTCOMES:
Arterial pressure | during procedure
anxiety | during and imediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, MD, PhD, Principal Investigator — University of Sao Paulo Medical School - FMUSP
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil